CLINICAL TRIAL: NCT02090881
Title: Comparison of a Portable and Non-Portable Ultrasound Machine in the Evaluation of Children With Sickle Cell Disease - A Pilot Study
Brief Title: Measurement of Cerebral Blood Flow Using Transcranial Doppler Ultrasound in Children With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13HH0858
Record Dates: First submitted 2013-10-31; First posted 2014-03-18 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound scan in ages 2-16 years (Experimental): Children aged 2-16 years of age with Sickle Cell Disease and under the care of consultant haematologist as part of the NHS screening programme.
  Interventions: Other: Ultrasound scan

INTERVENTIONS:
Other: Ultrasound scan — Trans cranial Doppler ultrasound examination of cerebral arterial blood flow

SUMMARY:
Sickle cell disease (SCD) affects haemoglobin - the molecule in blood cells which carries oxygen. It causes red blood cells to become abnormal crescent (or sickle)- shaped. Sickled red blood cells cannot travel through small blood vessels as easily as normal red blood cells which can lead to blockages. This means that oxygen may be prevented from getting to where it is needed. Individuals with sickle cell disease also suffer form abnormality in the lining of their blood vessels, which contributes to the damage.

Damage and blockage can occur in the blood vessels in the brain and means that children with sickle cell disease have a significant risk of suffering from strokes. Research has shown that transcranial Doppler ultrasonography can be used in this setting to identify children at most risk of getting strokes.

Ultrasound is therefore used in children with sickle cell disease to measure the blood flow in the vessels in the brain. This research has formed the basis of the National Health Service (NHS) Standard of Care for Sickle Cell Disease in the United Kingdom (UK) which uses transcranial Doppler ultrasonography at once a year to screen children with sickle cell disease aged 2 to 16.

Ultrasound is used because it is portable, does not uses ionising radiation such as x-rays, is non-invasive and gives good results. However, the results are dependent on the operator. This means that the screening service is provided by centres of excellence with experienced scanning staff visiting clinics in smaller hospitals with portable machines. There is a lack of research comparing the use of portable machines to laboratory-based machines. This is important because screening can identify children at high risk of stroke and may be used by clinical staff to make a decision about the care of the child.

DETAILED DESCRIPTION:
Please see above

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Sickle Cell Disease
* Under surveillance as part of the NHS Sickle Cell & Thalassaemia Screening Programme
* Children between the ages of 2 - 16 years old. Those under 16 years of age must be accompanied by a responsible adult.

Exclusion Criteria:

* Participants older than 16 years of age as this is outside the scope of the sickle cell screening programme.
* Individuals unable to give fully informed and voluntary consent.
* Individuals with inadequate temporal windows as it will not be possible to record measurements of velocity.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aslam, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Scan in Ages 2-16 Years
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound Scan in Ages 2-16 Years
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Time Average Mean of the Maximum (TAMM) in cm/Sec in Cerebral Arteries Using 2 Different Ultrasound Machines.
Description: A flow phantom was used to compare Time average mean maximum velocity measurements from a Philips IU-22 and Zonare Z-One ultrasound machine. 25 children with SCD (aged 2-15 years) attending the outpatient clinic at St. Mary's Hospital, Imperial College Healthcare NHS Trust as part of the NHS Sickle Cell & Thalassaemia (SC&T) screening programme, were studied. The Time Averaged Mean of the Maximum (TAMM) velocities in the middle cerebral artery (MCA) and stroke risk categorisation using the two ultrasound machines were compared.
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: cm/sec
Arm/Group | Ultrasound Scan in Ages 2-16 Years
Number analyzed (Participants) | 25
cm/sec
  Philips IU-22 | 120 [102 to 130]
  Zonare Z-One | 120 [102 to 130]

ADVERSE EVENTS:
Time Frame: 4 months period
Arm/Group | Ultrasound Scan in Ages 2-16 Years
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02090881/Prot_SAP_000.pdf